CLINICAL TRIAL: NCT04674124
Title: Feasibility and Acceptability of an Online Mindfulness-based Intervention for Mothers Within the Postpartum Period
Brief Title: Evaluation of an Online Mindfulness-based Course for New Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPID1920-0332
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: New Mothers Well-being; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Mindfulness Course (Experimental): Participants will be enrolled on a 9 week online mindfulness course.
  Interventions: Behavioral: Brief Online Mindfulness Intervention
- Delayed course materials (No Intervention): Participants will have access to the course materials at the closure of their involvement in the study.

INTERVENTIONS:
Behavioral: Brief Online Mindfulness Intervention — A nine-week mindfulness course compromising of 9x weekly 15 minute group sessions which will be on an online platform and daily micro meditations for participants to undertake.
  Other Names: 10ofZen
  Arms: Online Mindfulness Course

SUMMARY:
This research study is aiming to explore whether an online mindfulness programme is accessible and supportive for first time mothers who has a child who is less than 12 months old.

DETAILED DESCRIPTION:
This study is a randomised controlled trial (RCT) comparing an online mindfulness based course (10ofZen) with a treatment as usual group (delayed 10ofZen course materials). Participants will be informed about the study and asked to undertake a screening questionnaire to ensure the eligibility criteria is met. Following this, participants will be invited to give online consent. A battery of self-report measures will be administered online at baseline (week 0), post-intervention (week 10) and at follow-up (week 14). A sleep measure will also be undertaken and used as a co-variate during data analysis. At the end of participation in the research study, all participants will gain access to the course materials, including audio recordings of meditations and any written materials used within the course.

ELIGIBILITY:
Inclusion Criteria:

* Women who identify as a mother (Biological, adoptive, foster-carer or step-mum)
* Have an infant under the age of 12 months at baseline measures
* Sufficient English reading and listening abilities
* Access to the internet via an electronic device (phone, tablet, laptop or computer)
* Access to a mobile phone
* No prior experience of parenting a baby (under 12 months of age)

Exclusion Criteria:

* Previous completion of a formal 8-week mindfulness course or current mindfulness/meditation practice
* Currently pregnant
* Severe levels of depression and/or anxiety as measured by 15+ point on the Generalised Anxiety Disorder-7 and Patient Health Questionnaire-9 (NICE, 2011).
* Suicidal ideation or thoughts of self-harm in the last two weeks
* Currently experiencing symptoms of psychosis
* Diagnosis of Post Traumatic Stress Disorder (PTSD)
* Bereavement within the last six months which they still feel affected by.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who identify as a mother (Biological, adoptive, foster-carer or step-mum)
Enrollment: 112 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Differences in scores between groups at post intervention (10) and follow up (14) on the Short Warwick-Edinburgh Mental Well-Being Scale | Post-intervention and follow up ( i.e 10 & 14 weeks post baseline)
  Self-report measure of perceived well-being. Scores can range from 0-35. Higher scores are indicative of higher levels of subjective wellbeing.

SECONDARY OUTCOMES:
Differences in scores between groups at post intervention (10) and follow up (14) on the Maternal Postnatal Attachment Scale | Post-intervention ( i.e 10 & 14 weeks post baseline)
  Self-report measure of maternal emotional bond to the infant. Scores range from 0-95. Higher scores are indicative of higher levels of maternal emotional attachment.
Differences in scores between groups at post intervention (10) and follow up (14) on the Depression Anxiety Stress Scale - 21 | Post-intervention ( i.e 10 & 14 weeks post baseline)
  Self-report measure of depression, anxiety and stress. Scores range from 0-63 with higher scores being indicative of higher levels of depression, anxiety and/or stress.
Differences in scores between groups at post intervention (10) and follow up (14) Five Facet Mindfulness Questionnaire - 15 | Post-intervention ( i.e 10 & 14 weeks post baseline)
  Self-report measure of mindfulness traits. Scores can range between 15-75 with higher scores being indicative of higher levels of mindfulness traits.
Differences in scores between groups at post intervention (10) and follow up (14) on sleep quality | Post-intervention ( i.e 10 & 14 weeks post baseline)
  Self report measures on sleep quality ranging from 0 (very poor) to 10 (excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Pitman, BSc, MRes, Principal Investigator — Canterbury Christ Church University
Locations (1):
- Canterbury Christ Church University, Royal Tunbridge Wells, United Kingdom

IPD SHARING:
Plan to Share IPD: No